CLINICAL TRIAL: NCT06151795
Title: A Phase I Study to Evaluate the Safety, Biodistribution, Radiation Dosimetry, and Pharmacokinetics of XTR006 in Healthy Chinese Volunteers
Brief Title: A Study to Evaluate XTR006 in Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sinotau Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STB-XTR006-101
Record Dates: First submitted 2023-10-07; First posted 2023-11-30 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XTR006 (Experimental): Single dose 8.0-10.0 mCi intravenous injection of XTR006
  Interventions: Diagnostic Test: XTR006

INTERVENTIONS:
Diagnostic Test: XTR006 — Single dose intravenous injection of XTR006. Serial whole-body PET scan will be obtain after injection, blood and urine collection after injection for the assessment of pharmacokinetics.

SUMMARY:
XTR006 is a 18F-labeled positron emission tomography （PET）tracer for imaging tau protein in the brain. This phase I study investigated the safety, biodistribution, radiation dosimetry and Pharmacokinetics of XTR006 in 10 healthy elderly Chinese volunteers.

DETAILED DESCRIPTION:
XTR006 is a 18F-labeled PET tracer, for the quantification of neurofibrillary tangle (NFT) deposition in the brain. Brain NFT deposition is a pathologic finding in Alzheimer's Disease (AD), with brain NFT density shown to correlate with the severity of cognitive impairment in AD. This Phase I study will be open-labeled, nonrandomized, single center study. Enrolled 10 healthy elderly Chinese volunteers who meet all of the inclusion and none of the exclusion criteria. Subjects will receive 8-10mCi of XTR006 via IV injection. Safety and tolerability will be observed. Biodistribution, pharmacokinetics, and dosimetry will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between 50-70 years (included 50 & 70 years old) will be included;
2. Healthy or without serious diseases evaluated by the investigator based on the followings: medical history, vital signs, physical examination, electrocardiogram and clinical laboratory test results;
3. Electroencephalogram（EEG）examination result is "normal";
4. Aβ PET imaging is negative;
5. Mini-Mental State Examination (MMSE) score ≥ 28;
6. Normal routine blood and urine examination, liver function test, renal function test, biochemical test of serum troponin T and myocardial enzymes, or the abnormality of any test with no clinical significance;
7. Female subjects must take effective contraceptive measures during the study period and within 6 months after the last visit (effective contraceptive measures include sterilization, intrauterine hormone devices, condoms, contraceptives/agents, abstinence or partner removal of the vas deferens, etc.). Male subjects should agree to take contraception during the study period and within 6 months after the last visit;
8. Sign the informed consent form.

Exclusion Criteria:

1. Any previously diagnosed brain disease, such as cerebrovascular disease, inflammatory or infectious disease or any neurodegenerative disease, including any history of Parkinson's disease by physical or imaging manifestations, or history of traumatic brain injury, history of brain surgery or cranial internal hematoma by permanent brain injury;
2. Any history of severe diseases or undergoing unstable disease (such as unstable angina pectoris, dilated or hypertrophic cardiomyopathy, valvular heart disease, congenital heart disease, myocardial infarction, heart failure, chronic renal failure, chronic liver disease, severe lung disease, blood disease, diabetes, chronic infection, epilepsy, or mental illness);
3. The result of cranial magnetic resonance imaging (MRI) met the following imaging criteria: ① More than two infarct regions (diameter greater than 2 cm) outside the brain stem. ② Critical lacunar infarction, such as thalamus, hippocampus, entorhinal cortex and angular gyrus. ③ Fazekas score of high white matter damage ≥ 3 or minor axis of enlarged perivascular space (EPVS) > 3 mm determined by MRI examination;
4. Family history of dementia;
5. Medication in the past week or at the present that may interfere the result of clinical trial evaluated by the investigator;
6. Human immunodeficiency virus (HIV) hepatitis C or past test result of treponema pallidum antibody is positive, or hepatitis B surface antigen is positive;
7. History of coagulation disease or present coagulation disorder;
8. History of liver or gastrointestinal diseases or other conditions that can interfere the drug absorption, distribution, excretion or metabolism evaluated by the investigator;
9. Tumor history;
10. High risk of drug allergy (such as allergic asthma patients) or history of severe reactions to allergens;
11. Hyperreactive to alcohol;
12. History of alcohol or drug abuse;
13. Significant occupational exposure to ionizing radiation (e.g. more than 50 mSv/year), exposure to radioactive substances, ionizing radiation for therapeutic or research purposes in the past 10 years;
14. Completion of any medicine or treatments that may cause serious side effects or interfere the clinical trial's data evaluated by the investigator;
15. Participating other drug's clinical trial within 30 days before the enrollment;
16. Pregnant or lactating female;
17. Hospitalization due to illness during the screening period;
18. Other inappropriateness to the trial evaluated by the investigator.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events. | up to 7 days post injection.
  Safety Observation: Number of participants with adverse events and severe adverse events after drug injection.

SECONDARY OUTCOMES:
XTR006 Whole Body Effective Dose; | up to 5 hours
  Radiation dose estimates measured in millisieverts per megabecquerel (mSv/MBq) for the whole body obtained from Organ Level Internal radiation dosimetry code.

CONTACTS AND LOCATIONS:
Overall Officials: jianjun jia, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No